CLINICAL TRIAL: NCT06197477
Title: Development of Novel Assessments for Indoor Air Quality Monitoring and Impact on Children's Health - Cohorts in Schools & Biomarkers of Exposure
Brief Title: Indoor Air Quality Monitoring and Impact on Children's Health
Acronym: LEARN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Tim Nawrot, Professor, Hasselt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Hasselt University
Record Dates: First submitted 2023-09-28; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Cognition
Keywords: indoor air pollution; indoor air quality; cognition in children

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air purification (Experimental): The intervention will consist of air purification placed in the classrooms.
  Interventions: Device: OurAir SQ 1750 - Mobile Air Purification System for indoor
- Control (Sham Comparator): Filtration will be turned off in the air purifier placed in the classrooms in the control part of the study.
  Interventions: Device: Sham intervention

INTERVENTIONS:
Device: OurAir SQ 1750 - Mobile Air Purification System for indoor — Filtration device will be placed in classrooms. Computational Fluid Dynamics simulations will be used to find optimal position and operation mode for air purification systems in classrooms.
  Arms: Air purification
Device: Sham intervention — Filtration will be turned off in the control part of the study and then will be turned on during the intervention.
  Arms: Control

SUMMARY:
This study aims at understanding the relation between indoor air quality in schools, including both chemical and microbiological determinants, and cognition in children by gathering data across different parts of Europe

DETAILED DESCRIPTION:
The LEARN project, funded by the European Commission, aims to gain an in-depth understanding about indoor air quality in schools and its impact on children's cognitive development. This involves evaluating school cohorts in three different countries (Belgium, Greece and Denmark). In participating schools, we measure and characterise indoor and outdoor air pollutants and evaluate the presence of exposure biomarkers and their effect on children's cognition. Measuring indoor air quality, exposure and creating remedial strategies are crucial steps to improve air quality in the school environment and ensure the well-being of children.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls
* Attending school in the 4th -6th grade in elementary schools included in the study
* Signed informed consent form by legal representative

Exclusion Criteria:

* Insufficient knowledge of local language (ie. Dutch, Greek, Danish) by child or parents

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Correct Detection of continuous Performance Test | at the end of the intervention and at the end of the sham intervention
  Change in the number of times the child responded correctly to the target alphanumeric stimulus. Higher rates of correct detections indicate better attentional capacity.
Change in the number of correct substitutions of Symbol Digit Modalities Test | at the end of the intervention and at the end of the sham intervention
  Change in the the number of correct substitutions the child performed. Higher number of correct substitutions indicate better information processing ability.
Change in the Memory Span Task score | at the end of the intervention and at the end of the sham intervention
  Change in the number of longest list of items that a child can repeat back in correct order. Longer list of recalled items indicate better short term memory
Change in the Signal Detection Test score | at the end of the intervention and at the end of the sham intervention
  Change in the number of correct detection of signals. Higher rates of correct detection indicate better perception ability

CONTACTS AND LOCATIONS:
Overall Officials: Tim Nawrot, PhD, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Belgium

IPD SHARING:
Plan to Share IPD: No